CLINICAL TRIAL: NCT01531478
Title: Long-term Follow-up of Childhood Cancer Survivors in the Rhône-Alpes and Auvergne Regions of France
Acronym: SALTO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1008102; 2010-A00853-36 (Other: AFSSAPS)
Record Dates: First submitted 2011-07-20; First posted 2012-02-13 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Cancer; Sequels; Complications
Keywords: Childhood cancer; Cancer; Sequels; Complications; Chemotherapy; Radiotherapy; Surgery
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Young adult survivors of childhood cancer: Young adult survivors of childhood cancer diagnosed between 1987 and 1992 in the Rhône-Alpes and Auvergne regions of France.
  Interventions: Other: Unique medical visit of the study

INTERVENTIONS:
Other: Unique medical visit of the study — The visit will be with an oncologist specialized in the long-term follow-up of cured pediatric cancer patients. The examination will consist in weight and height measurements, a clinical examination and a measurement of arterial pressure. The list of drugs taken in the last two years, as well as all health issues encountered since the cancer treatment, will be collected. Success in education, career and, family status will also be discussed.
  After the medical examination, patients will be offered a visit with a psychologist in order to assess their psychopathological outcomes. This questionnaire is a interquestionnaire designed to screen axis I psychopathological conditions. It includes an evaluation of all types of risk-taking behavior (alcohol, drugs, anorexia and bulimia).

SUMMARY:
Childhood cancers are rare, and today 75% of patients survive them. An estimated one out of 850 French persons has survived childhood cancer. However, the complications of chemotherapy, radiotherapy or surgery can lead to a higher risk of secondary mortality, which the literature estimates is at 14%. Regular care has a positive impact on the quality of life and health of adults who survived cancer during their childhoods. It aims to detect the potential long-lasting effects of cancer and to provide therapeutic education and psychological care. Thanks to cancer registries, several countries (USA, Canada, UK, Germany, the Netherlands) have developed long-term care structures which function with specially trained adult medicine practitioners. There are only two structures in France: the Long-Term Oncology/Hematology Follow-Up Clinic, headed by Dr François Pein, in Nantes (France), and the LEA program for the follow-up of children treated for leukemia in the PACA-Corse and Lorraine regions of France, which began in 2003 and has since been extended to other centers.

The Rhône-Alpes and Auvergne regions have had childhood cancer registries since 1987; they compile about 200 new cases a year. The Rhône-Alpes registry has conducted a preliminary trial on children (0-15 years old) diagnosed with cancer between 1987 and 1992. They analyzed the correlation between patients' quality of life and the long-term medical effect of cancer and treatment, both recorded in patients' medical files and declared by patients. These young adults who survived pediatric cancer appear to suffer from and declare many complications, although this does not impact their global quality of life much. There is a negative correlation between the number of complications (observed or declared) and the global quality of life score, but only three types of complications play a significant role (motor function complications, auditory complications, and alopecia.) In addition, there is a significant mismatch between patients's perceived health (what they say they experience), and the information contained in their medical files. These young adults expressed the need for their impressions to be better taken into account by health care professionals. This study does not assess patients' psychopathological characteristics.

DETAILED DESCRIPTION:
Results will help identify long-term complications, respond to patients' expectations, and evaluate the feasibility of conducting such a follow-up in all patients. They should guide the choice of the most appropriate tools for care, help assess needs in terms of collaboration with adult care staff, and identify potential partners.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with cancer between 01/01/1987 and 31/12/1992, before age 15, and living in Auvergne or Rhône-Alpes (France)
* Being a beneficiary of health insurance
* Having signed the informed consent form

Exclusion Criteria:

* Having been diagnosed with leukemia as a primary cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective cohort study in non-leukemia cancer survivors diagnosed between 1987 and 1992 in the Rhône-Alpes and Auvergne regions of France, who were younger than 15 years at the time of diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2011-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Medical complications (post cancer treatment) | 15 years after the end of the cancer treatment
  The investigators note the medical complications from the end of their cancer treatment to the inclusion visit. Theses complications depend on the type of treatment received.

SECONDARY OUTCOMES:
MINI questionnaire score | 15 years after the end of the cancer treatment
  The investigators measured the psychological complications (post cancer treatment) by MINI questionnaire score.

CONTACTS AND LOCATIONS:
Overall Officials: Claire BERGER, MD, Principal Investigator — CHU de Saint-Etienne
Locations (4):
- France (4):
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de Grenoble, Grenoble
  - IHOP, Lyon
  - CHU de Saint-Etienne, Saint-Etienne

REFERENCES:
- [Derived] Tardy F, Casagranda L, Protiere A, Buisson-Papet G, Garcin A, Trombert-Paviot B, Freycon C, Marec-Berard P, Massoubre C, Berger C. Long-Term Clinical and Psychiatric Complications of Young Adults Cured of a Pediatric Bone Tumor Diagnosed Between 1987 and 1999 in Rhone: Alpes Region (France). J Adolesc Young Adult Oncol. 2022 Dec;11(6):571-579. doi: 10.1089/jayao.2021.0145. Epub 2022 Jan 18. PMID 35049375